CLINICAL TRIAL: NCT04809948
Title: Impact of COVID 19 Vaccine on Safety, Blood Elements, and Immunogenicity of the Egyptian Population
Brief Title: Effects of COVID 19 Vaccine on Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, lecturer, Assiut University
Other Study IDs: COVID 19 Vaccine
Record Dates: First submitted 2021-03-14; First posted 2021-03-22 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: COVID 19 Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Biological: viral vector vaccine — AstraZeneca vaccine

SUMMARY:
The aim of this study is to identify adverse events following vaccination by the COVID-19 vaccine by evaluating adverse side effects, hematological values; immunogenicity in the Egyptian candidates in response to COVID-19 vaccine, summarizing the which may occur following administration of COVID-19 vaccine.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an emerging respiratory infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that had infected more than 100 million individuals and caused more than 2 million deaths worldwide by February 13, 2021. A safe and effective vaccination trials against COVID-19 is urgently needed. There are currently more than 160 COVID-19 candidate vaccines in development worldwide, and 25 are in different phases of clinical trials using different platforms.

The efficacy and immunogenicity of vaccines varies depending on the study cohort. Race and ethnicity were shown to affect the antibody responses to the rubella vaccine, which elicited significantly higher titers in children of African ethnicity compared to those of European descent or Hispanic ethnicity, likely, disparities in serologic responses to vaccines were also observed between different ethnic groups for the Haemophilus influenzae type b-tetanus toxoid conjugate vaccine , or the Haemophilus influenzae type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine . thus keeping the race an important factor in studding its effect on immunogenicity of vaccine. Thus keeping the race an important factor in studding its effect on immunogenicity of vaccine, which pushed us to estimate immunogenicity in Egyptian population after vaccination with the inactivated COVID-19 vaccine.

Heamatological changes after vaccination had been detected in many researches; lecuocytosis was found shortly after vaccination of infants, which was primarily a neutrophilia but no participant received antibiotics and all remained well at follow-up . In a case series study, also leukocytosis with fever was detected following pneumococcal vaccine administration . On the other hand, neutropenia was detected following a new vaccine against Shigella sonnei . Platelets abnormalities also had been detected following vaccination, a previous example is idiopathic thrombocytopenic purpura, linked to the administration of measles-containing vaccines .

ELIGIBILITY:
Inclusion Criteria:

1. People aged 18-80 years.
2. Negative for serum-specific IgM/IgG antibodies against SARS-CoV-2, as measured by a commercial kit (Innovita, China) at the time of screening.

Exclusion Criteria:

1. A history of infection with SARS-CoV 3 months before the vaccine.
2. Fever, cough, runny nose, sore throat, diarrhoea, dyspnoea, or tachypnoea in the 14 days before vaccination.
3. Pregnancy.
4. A history of seizures or mental illness.
5. Being on immunosuppressive agents.
6. Being on anticoagulation therapy.
7. Being unable to comply with the study schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HCWs in Assiut University Hospitals accepted to take vaccine
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
serological antibodies against SARS-CoV-2 e | change from baseline at one month after first dose
  Total IgG titer
serological antibodies against SARS-CoV-2 e | one month after second dose
  Total IgG titer
Complete blood count (CBC) | change from baseline at one month after first dose
  to evaluate total leucocyte count TLC
Complete blood count (CBC) | one month after second dose
  to evaluate total leucocyte count TLC
Complete blood count (CBC) | change from baseline at one month after first dose
  absolute neutrophilic count (ANC)
Complete blood count (CBC) | one month after second dose
  absolute neutrophilic count (ANC)
Complete blood count (CBC) | change from baseline at one month after first dose
  platelets (PLTs)
Complete blood count (CBC) | one month after second dose
  platelets (PLTs)
Complete blood count (CBC) | change from baseline at one month after first dose
  hemoglobin level
Complete blood count (CBC) | one month after second dose
  hemoglobin level
Adverse clinical symptoms after vaccine | up to one week after first dose
  asking about possible recorded side effects as
  * Local: irritation, erythema, swelling, or itching.
  * Systemic: headache, dizziness, difficult sleep, flush, muscle pain, joint pain, fatigue, fever, chills, sore throat, nasal congestion, nasal bleeds, sneezing, runny nose, cough, dyspnoea, palpitation, nausea, vomiting, diarrhoea, constipation, stomach pain, loss of appetite, acute allergic reaction, acne, abnormal taste, loss of taste, mouth ulcers, toothache, ear pain, eye pain, and/or lymphadenopathy.

REFERENCES:
- [Background] Spinelli A, Pellino G. COVID-19 pandemic: perspectives on an unfolding crisis. Br J Surg. 2020 Jun;107(7):785-787. doi: 10.1002/bjs.11627. Epub 2020 Mar 23. No abstract available. PMID 32191340
- [Background] Stern PL. Key steps in vaccine development. Ann Allergy Asthma Immunol. 2020 Jul;125(1):17-27. doi: 10.1016/j.anai.2020.01.025. Epub 2020 Feb 7. PMID 32044451
- [Background] Xia S, Duan K, Zhang Y, Zhao D, Zhang H, Xie Z, Li X, Peng C, Zhang Y, Zhang W, Yang Y, Chen W, Gao X, You W, Wang X, Wang Z, Shi Z, Wang Y, Yang X, Zhang L, Huang L, Wang Q, Lu J, Yang Y, Guo J, Zhou W, Wan X, Wu C, Wang W, Huang S, Du J, Meng Z, Pan A, Yuan Z, Shen S, Guo W, Yang X. Effect of an Inactivated Vaccine Against SARS-CoV-2 on Safety and Immunogenicity Outcomes: Interim Analysis of 2 Randomized Clinical Trials. JAMA. 2020 Sep 8;324(10):951-960. doi: 10.1001/jama.2020.15543. PMID 32789505
- [Background] Haralambieva IH, Salk HM, Lambert ND, Ovsyannikova IG, Kennedy RB, Warner ND, Pankratz VS, Poland GA. Associations between race, sex and immune response variations to rubella vaccination in two independent cohorts. Vaccine. 2014 Apr 7;32(17):1946-53. doi: 10.1016/j.vaccine.2014.01.090. Epub 2014 Feb 13. PMID 24530932
- [Background] Prentice S, Kamushaaga Z, Nash SB, Elliott AM, Dockrell HM, Cose S. Post-immunization leucocytosis and its implications for the management of febrile infants. Vaccine. 2018 May 11;36(20):2870-2875. doi: 10.1016/j.vaccine.2018.03.026. Epub 2018 Apr 11. PMID 29655624
- [Background] von Elten KA, Duran LL, Banks TA, Banks TA, Collins LC, Collins LC. Systemic inflammatory reaction after pneumococcal vaccine: a case series. Hum Vaccin Immunother. 2014;10(6):1767-70. doi: 10.4161/hv.28559. Epub 2014 Mar 18. PMID 24642659
- [Background] Muturi-Kioi V, Lewis D, Launay O, Leroux-Roels G, Anemona A, Loulergue P, Bodinham CL, Aerssens A, Groth N, Saul A, Podda A. Neutropenia as an Adverse Event following Vaccination: Results from Randomized Clinical Trials in Healthy Adults and Systematic Review. PLoS One. 2016 Aug 4;11(8):e0157385. doi: 10.1371/journal.pone.0157385. eCollection 2016. PMID 27490698